CLINICAL TRIAL: NCT06080672
Title: The Effect of Disclosing Dental Plaque on Plaque Index and Gingival Index in Istanbul Medipol University Faculty of Dentistry Students
Brief Title: The Effect of Disclosing Dental Plaque on Plaque Index and Gingival Index in Faculty of Dentistry Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nilüfer Üstün, associate professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-2361
Record Dates: First submitted 2023-09-20; First posted 2023-10-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Indexes; Oral Health
Keywords: Dental students; Plaque index; Gingival index; Plaque disclosing agents

STUDY DESIGN:
Intervention Model Description: Group 1: Students, whose first records (plaque index, gingival index) are taken after the examination by the periodontology specialist, will be taught how to brush their teeth with the Modified Bass Technique and how to use dental floss/interdental brush. Students will then be asked to brush their teeth.
  Group 2: The students, whose initial records (plaque index, gingival index) are taken after the examination by the periodontology specialist, will be taught how to brush their teeth with the Modified Bass Technique and how to use dental floss/interdental brush. After staining the teeth with a plaque disclosing agent, they will be shown in the mirror. Then the students will then be asked to brush their teeth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (dental examination-training-tooth brushing) (Experimental): Students, whose first records (plaque index, gingival index) are taken after the examination by the periodontology specialist, will be taught how to brush their teeth with the Modified Bass Technique and how to use dental floss/interdental brush. Students will then be asked to brush their teeth.
  Interventions: Other: Experimental: Group 1 (dental examination-training-tooth brushing) Experimental: Group 2 (dental examination-training-plaque disclosing-tooth brushing)
- Group 2 (dental examination-training-plaque disclosing-tooth brushing) (Experimental): The students, whose initial records (plaque index, gingival index) are taken after the examination by the periodontology specialist, will be taught how to brush their teeth with the Modified Bass Technique and how to use dental floss/interdental brush. After staining the teeth with a plaque disclosing agent, they will be shown in the mirror. Then the students will then be asked to brush their teeth.
  Interventions: Other: Experimental: Group 1 (dental examination-training-tooth brushing) Experimental: Group 2 (dental examination-training-plaque disclosing-tooth brushing)

INTERVENTIONS:
Other: Experimental: Group 1 (dental examination-training-tooth brushing) Experimental: Group 2 (dental examination-training-plaque disclosing-tooth brushing) — All participants will be examined and their decay, filling and extracted teeth, plaque index and gingival index measurements will be recorded. Plaque disclosing will be applied to Group 2 after brushing training.

SUMMARY:
The hypothesis of this study is; using the tooth disclosing agents by individuals has a positive effect on oral care and as if it is an effective method in improving oral health. Therefore, the aim of this study is to assess the effect of visual guidance of plaque disclosing agents on plaque removal efficacy for patients versus the group of patients evaluated without any tools.

Istanbul Medipol University Faculty of Dentistry 4th grade students are going to be invited to the study. The study will carry out with a total of 124 students. The students who are systemically healthy, drug-free, and at least 20 teeth in the mouth will be included in the study. Smokers, those undergoing orthodontic treatment, the presence of pain or infection that may prevent brushing, pregnant/breastfeeding students, and students who do not agree to participate in the study will not include to the study.

After the initial records (Plaque index and Gingival Index and DMFT- caries, missing teeth due to caries, filled teeth) were obtained, the students in the study will randomly divide into 2 groups:

Group 1; Control Group (n=62) After explaining the Modified Bass Technique and the use of dental floss/interface brush, students will be asked to brush their teeth.

Group 2; Test Group (n=62) After explaining the Modified Bass Technique and the use of dental floss/interface brush, the teeth will stain with a plaque disclosing agent, the plaque is going to be shown in the mirror and then the students will brush their teeth.

Post-operatively, periodontal parameters will be evaluated. Plaque index and gingival index will be measured immediately after brushing, 1 week, 1 months are going to be compared to baseline. A single investigator will make measurements of Gingival Index (GI, Löe and Sillness-1967) and Plaque Index (PI, Sillness and Löe-1964) using a Williams periodontal probe. Measurements will be obtained from 4 surfaces of all teeth (mesiobuccal, midbuccal, distobuccal, midlingual) except third molar teeth, and the values obtained will be summed and averaged, and the average of one tooth. Then, these values will be summed up and averaged, and the mean PI and GI of the individual will be obtained. The outcomes of the two groups will be evaluated by statistical analysis.

DETAILED DESCRIPTION:
The study will be carried out in Istanbul Medipol University Department of Pedodontics, period between October 2023- January 2024. Ethical approval for the study was received from Istanbul Medipol University Ethics Committee. (REF: E-10840098-772.02-2361). The students who agreed to participate in the study will be informed about the study and the written informed consents will be obtained from all participants included in the study.

At the end of the study, 124 students whose measurements were completed will be included in the research. A randomization list was generated using online software (http://www.graphpad.com/quickcalcs/index.cfm), where students enrolled on the study were randomized into 2 groups with an allocation ratio of 1:1. The random allocation sequence was generated by an independent researcher; thus, the operator and observer were blinded to the assignment of the study participants to the groups as follows:

Group 1: Students, whose first records (plaque index, gingival index) are taken after the examination by the periodontology specialist, will be taught how to brush their teeth with the Modified Bass Technique and how to use dental floss/interdental brush. Students will then be asked to brush their teeth.

Group 2: The students, whose initial records (plaque index, gingival index) are taken after the examination by the periodontology specialist, will be taught how to brush their teeth with the Modified Bass Technique and how to use dental floss/interdental brush. After staining the teeth with a plaque disclosing agent, they will be shown in the mirror. Then the students will then be asked to brush their teeth.

Study Design This randomized clinical study will last in three months. According to data from the previous studies, the desired sample size (n=124) was calculated. Among the 204 students who were examined in the beginning, 124 students who met the inclusion criteria will be included in the study to be protected from dropouts.

In the beginning, students are going to fill out an examination form consisting of questions about attitudes of their oral and dental health and the demographic data of the study group. Examination forms consisted of; name-surname, birthdate, examination date, gender, tooth brushing habits (yes or no, and how often they brush their teeth), the use of dental floss and/or an interdental (interface) brush, and how often they use them, the use of mouthwash and/or mouth spray, the last time of they visited a dentist, bleeding of their gums (yes/no). Then, the students will be examined and their DMFT index (decayed, filled, and missing teeth), baseline plaque index and gingival index measurements will be recorded. The students will randomly divide into two groups. All students will be trained about toothbrushing by Modified Bass Technique and the use of dental floss/interface brush by the video presentation and demonstrating with models from the same instructer. Commercially available standard toothpastes will be distributed to students. The students in the control group will be asked to brush their teeth with the technique taught. The teeth of the students in the second group, which is the test group, to stain the teeth Mira 2-tone Solution (Hager&Werken) will be used to visualize dental plaque. After the staining, the students will rinse their mouths with water and the stained tooth surfaces will be shown with the help of hand mirrors. Then the second groups students will brush their teeth with Modified Bass Technique and only the plaque index will be measured again. One week later, the students will be called for control again, and plaque index and gingival index measurements will be repeated in the test group after plaque disclosing and in the control group without disclosing. At the end of one month, the measurements will be repeated in both groups and the data will be recorded.

Gingival Index (GI, Löe and Sillness-1967) and Plaque Index (PI, Sillness and Löe-1964) measurements will be done by a single investigator using a Williams periodontal probe. Measurements will be obtained from 4 surfaces of all teeth (mesiobuccal, midbuccal, distobuccal, midlingual) except third molars, and the values obtained will be summed and averaged, and the average of one tooth; Then, these values will be summed up and averaged, and the mean PI and GI of the individual will be obtained.

The distribution of variables will be analyzed using the Kolmogorov-Smirnov test. Student's t-test and chi-square test will be used to compare the quantitative and qualitative data of the two groups. Spearman's correlation coefficient (R) will be used to evaluate relationships between periodontal status data (PI, GI, DMFT).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Being drug-free
* Have at least twenty teeth in the mouth

Exclusion Criteria:

* Smokers
* Undergoing orthodontic treatment
* Has pain or infection that prevent brushing
* Pregnant/breastfeeding

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Filling examination forms | The first 10 minutes of the first visit
  The form containing questions about the study group's attitudes towards oral and dental health and their demographic data is filled out by the participants.
Dental examination | Immediately after the students filled the examination forms at the first visit
  Oral and dental examination will be done by a specialist periodontist, and DMFT index (total number of decayed, filled, and missing teeth) will be recorded
Plaque Index (PI, Sillness and Löe-1964) measurements | During the dental examination procedure
  Measurements will be done by a single investigator using a Williams periodontal probe. Measurements will be obtained from 4 surfaces of all teeth (mesiobuccal, midbuccal, distobuccal, midlingual) except third molars, and the values obtained will be summed and averaged, and the average of one tooth; Then, these values will be summed up and averaged, and the mean PI of the individual will be obtained. The PI which is going to be used to determine the oral hygiene level of the individuals included in the study will be evaluated as follows:
  0: No bacterial plaque on the tooth surface.
  1. There is plaque in the form of film and can be seen with the help of a probe.
  2. There is moderate soft attachment visible to the naked eye.
  3. There is a visible dense soft appendage filling the gingival sulcus on the tooth surface.
Gingival Index (GI, Löe and Sillness-1967) measurements | During the dental examination procedure
  Measurements will be done by a single investigator using a Williams periodontal probe. Measurements will be obtained from 4 surfaces of all teeth (mesiobuccal, midbuccal, distobuccal, midlingual) except third molars, and the values obtained will be summed and averaged, and the average of one tooth; Then, these values will be summed up and averaged, and the mean GI of the individual will be obtained.
  GI will be evaluated according to the following criteria:
  0: Healthy gingiva.
  1. There is mild inflammation, discoloration and edema, no bleeding on probing.
  2. Moderate inflammation, marked redness, edema, and bleeding on probing.
  3. Severe inflammation, prominent redness and edema, ulceration, spontaneous bleeding tendency.
Green and Vermillion Oral Hygiene Index-Simplified | 30th minute of the first visit
  In the second group, to stain the teeth Mira 2-tone Solution (Hager&Werken) will be used to visualize dental plaque. The amount of plaque will be measured by staining method from different surfaces of six teeth, two from the front area and four from the back area. 2 drops of Mira-2-tone plaque staining solution will be placed in plastic containers and be applied to the teeth with a brush. Measurements will be done from the buccal surfaces of teeth 16 and 26, the lingual surfaces of teeth 36 and 46, and the labial surfaces of teeth 11 and 31. The amount of plaque will be graded with 4 separate scores from 0 to 3, depending on the size of the surface area stained with the staining solution. The index will be calculated by dividing the total values by the number of surfaces.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Üstün, Ph.D., Principal Investigator — Medipol University; Beyza Ballı Akgöl, Ph.D., Principal Investigator — Antalya Bilim University; Merve Bayram, Ph.D., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Department of Pedodontics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng Y, Wu R, Qu W, Wu W, Chen J, Fang J, Chen Y, Farella M, Mei L. Effect of visual method vs plaque disclosure in enhancing oral hygiene in adolescents and young adults: a single-blind randomized controlled trial. Am J Orthod Dentofacial Orthop. 2014 Mar;145(3):280-6. doi: 10.1016/j.ajodo.2013.10.021. PMID 24582019
- [Background] da Silva CH, Paranhos Hde F. Efficacy of biofilm disclosing agent and of three brushes in the control of complete denture cleansing. J Appl Oral Sci. 2006 Dec;14(6):454-9. doi: 10.1590/s1678-77572006000600012. PMID 19089247
- [Background] Silva DD, Goncalo Cda S, Sousa Mda L, Wada RS. Aggregation of plaque disclosing agent in a dentifrice. J Appl Oral Sci. 2004 Jun;12(2):154-8. doi: 10.1590/s1678-77572004000200014. PMID 21365140
- [Background] Mensi M, Scotti E, Sordillo A, Agosti R, Calza S. Plaque disclosing agent as a guide for professional biofilm removal: A randomized controlled clinical trial. Int J Dent Hyg. 2020 Aug;18(3):285-294. doi: 10.1111/idh.12442. Epub 2020 May 26. PMID 32348624
- [Background] Montevecchi M, Checchi V, Gatto MR, Klein S, Checchi L. The use of a disclosing agent during resective periodontal surgery for improved removal of biofilm. Open Dent J. 2012;6:46-50. doi: 10.2174/1874210601206010046. Epub 2012 Feb 6. PMID 22371815